CLINICAL TRIAL: NCT00509886
Title: Non-prescription Versus Prescription Topical Treatments Versus no Treatment in the Control of Sweating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Murad Alam, MD, Northwestern University Dermatology department
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: STU00000722
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Hyperhidrosis; Excess Sweating
MeSH Terms: conditions — Hyperhidrosis | interventions — Aluminum Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ARMs were randomized. One side of the body received treatment with one antiperspirant and the contralateral side with a different antiperspirant.
  Interventions: Drug: Drysol
- 2 (Experimental): ARMs were randomized. One side of the body received treatment with one antiperspirant and the contralateral side with a different antiperspirant.
  Interventions: Drug: Drioff

INTERVENTIONS:
Drug: Drysol — 20% aluminum chloride hexahydrate
  Arms: 1
Drug: Drioff — 1% aluminum acetate
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effectiveness of the prescription treatment compared to the non-prescription treatment. It is hypothesized that the prescription treatment will have a significantly greater effect than the non-prescription treatment on decreasing excess sweating.

DETAILED DESCRIPTION:
The objective of this study is to assess the effectiveness of the prescription treatment compared to the non-prescription treatment. It is hypothesized that the prescription treatment will have a significantly greater effect than the non-prescription treatment on decreasing excess sweating.

ELIGIBILITY:
Inclusion Criteria:

* age 21-30 years
* males and females
* The subjects are in good health.
* The subjects have willingness and the ability to understand and provide informed consent for participation in the study.

Exclusion Criteria:

* Subjects with primary hyperhidrosis
* Subjects who are unable to withstand prolonged heat exposure or who have self-reported history of cardiovascular or respiratory disorders.
* Subjects who are unable to give informed consent.
* Subjects with mental illness.
* Subjects who are pregnant or nursing.
* Subjects with systemic or local skin disease and/or infection that may interfere with the conduct of the study.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Gravimetric analysis | 3 hours

SECONDARY OUTCOMES:
Subject sweat assessment | 3 hours
HDSS | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University dermatology; Dennis West, PhD, Study Director — Northwestern University dermatology
Locations (1):
- Northwestern University Dermatology, Chicago, Illinois, United States